CLINICAL TRIAL: NCT01411969
Title: Acoustic Rhinometry: Impact of External Nasal Dilator on the Two First Notches of the Rhinogram
Brief Title: Impact of External Nasal Dilator on the Rhinogram
Acronym: ARENDS
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Carlos Eduardo Nazareth Nigro, Ph.D, University of Sao Paulo General Hospital
Other Study IDs: 306/03
Record Dates: First submitted 2011-07-26; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-06

CONDITIONS: Nasal Obstruction
Keywords: external nasal dilator strip; nasal valve; acoustic rhinometry
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- External nasal dilator, decongestion
  Interventions: Drug: External Nasal Dilator Strip; 0.05% oxymetazoline chloride

INTERVENTIONS:
Drug: External Nasal Dilator Strip; 0.05% oxymetazoline chloride — External Nasal Dilator Strip placed above the upper lateral cartilage; 20 minutes after decongestion with 0.05% oxymetazoline chloride applied as an aerosol spray (two times); after decongestion with ENDS.
  Other Names: Breath Right®

SUMMARY:
The aim of this study is to present new data for a better understanding of the anatomic correlation of these two notches.

This study included 32 nasal cavities (16 individuals) with external nasal dilator strip (Breath Right®) and after decongestion (0.05% oxymetazoline chloride applied as an aerosol spray);

DETAILED DESCRIPTION:
Acoustic rhinometry is more accurate in the anterior portion of the nasal cavities, from the nostril to the nasal valve (NV), the most important site of nasal obstruction. Literature presents different opinions regarding the anatomical correlation of the two notches at the beginning of the rhinogram curve in normal adult Caucasian individuals.

This prospective study included 32 nasal cavities under the following conditions: 1st - basal condition; 2nd - with external nasal dilator strip (ENDS) (Breath Right®); 3rd - after decongestion (0.05% oxymetazoline chloride applied as an aerosol spray); 4th - after decongestion with ENDS.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Caucasian

Exclusion Criteria:

* Allergies, sinusitis, nasal polyps, external nasal deformities congenital or acquired, obstructive nasal deviation and regular use of any drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 32 nasal cavities of 16 normal adult Caucasian individuals
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao F Mello-Jr, Ph.D, Study Director — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Seren E. The effect of an adhesive external nasal dilator strip on the inspiratory nasal airflow. Am J Rhinol Allergy. 2010 Jan-Feb;24(1):e29-31. doi: 10.2500/ajra.2010.24.3426. PMID 20109318
- [Derived] Nigro CE, Mion O, Mello JF Jr, Voegels RL, Roithmann R. Acoustic rhinometry: impact of external nasal dilator on the two first notches of the rhinogram. Am J Rhinol Allergy. 2011 Nov-Dec;25(6):e247-50. doi: 10.2500/ajra.2011.25.3708. PMID 22185733